CLINICAL TRIAL: NCT01312376
Title: A Phase-1 Trial of Adoptive Transfer of Vaccine-Primed CD3/CD28-Costimulated Autologous T-Cells Combined With Vaccine Boost and Bevacizumab for Recurrent Ovarian Fallopian Tube or Primary Peritoneal Cancer Previously Vaccinated With Autologous Tumor Vaccine
Brief Title: Autologous T-Cells Combined With Autologous OC-DC Vaccine in Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 26810, R01 FD 003520; FDA 00PD (Other Grant/Funding Number: R01FD003520-04)
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Ovarian Carcinoma; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Bevacizumab; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: OC-DC vaccine — All subjects will receive a dose of 5-10 million cells of OC-DC intradermally
Drug: Bevacizumab — Patients will start receiving Bevacizumab at 15 mg/kg starting Day 30 and every 4 weeks thereafter until end of study.
Drug: cyclophosphamide 300 mg/m2/d for 3 days — All subjects will receive a single course of outpatient lympho-depleting chemotherapy with intravenous cyclophosphamide for 300 mg/m2/d for 3 days.
Drug: fludarabine 30 mg/m2/d for 3 days — All subjects will receive a single course of outpatient lympho-depleting chemotherapy with intravenous fludarabine 30 mg/m2/d for 3 days
Drug: ex vivo CD3/CD28-costimulated vaccine-primed peripheral blood autologous T cells — All subjects will receive a single intravenous infusion of ex vivo CD3/CD28-costimulated vaccine-primed peripheral blood autologous T-cells at the starting dose of 10-15 x 109 (10-15 billion) T-cells with escalating doses in cohort 2 and 3.

SUMMARY:
This is a phase-I clinical trial to determine the feasibility and safety of Cyclophosphamide/Fludarabine Lymphodepletion and an immunomodulatory combination of Interferon-alpha Bevacizumab and Aspirin followed by adoptive transfer of vaccine-primed ex vivo CD3/CD28-costimulated peripheral blood autologous T cells and vaccination with whole tumor vaccine administered intradermally in combination with Bevacizumab in patients with recurrent ovarian cancer fallopian tube or primary peritoneal cancer. (Funding Source - FDA OOPD)

DETAILED DESCRIPTION:
This is a phase-I clinical trial to determine the feasibility and safety of cyclophosphamide/fludarabine lymphodepletion and an immunomodulatory combination of Interferon-alpha (INF-a), Bevacizumab and Aspirin, followed by adoptive transfer of vaccine-primed, ex vivo CD3/CD28-costimulated peripheral blood autologous T-cells, and vaccination with whole tumor vaccine, administered intradermally in combination with Bevacizumab in patients with recurrent ovarian cancer, fallopian tube or primary peritoneal cancer who previously underwent induction vaccination with whole tumor vaccine.

Subjects will receive T-lymphocytes infusion at a dose of 20 billion ± 20% cells for all patients. Subjects who cant meet target dose level can still enroll but will be analyzed separately.

Before T-cell infusion, all subjects will undergo lymphodepletion with a single course of outpatient high-dose lymphodepleting chemotherapy with intravenous cyclophosphamide (300 mg/m2/d for 3 consecutive Days) and intravenous fludarabine (30 mg/m2/d for 3 consecutive Days on Days -5 to -3).

Subjects enrolled in this study will receive an immunomodulatory cycle of (Bevacizumab and Aspirin) ~14 Days before apheresis (if they do not have a frozen apheresis product from a previous collection) and another cycle between apheresis and T-cell infusion (approx. from Day -20 through Day -7, (+/- 5 Days)). The immunomodulatory cycle will consist of the following: intravenous 10 mg/kg Bevacizumab on Day -35, and Day -20 (+/- 5 Days), and 325 mg Enteric Coated Aspirin orally starting Day -35 for 14 Days and starting on Day -20 for 14 Days. They will also receive three subcutaneous injections of Interferon-alpha (Intron®a 2b) (INF-a) (subjects will have the option to self administer Interferon-alpha and they will be provided instructions) at a dose of 5 MIU on Days -3, -2 and -1. EX vivo CD3/CD28-costimulated lymphocytes will be infused ~1-2 Days after last Day of interferon-alpha treatment, ideally on Day 0.

All subjects will receive a dose of 5-10 million cells of OC-DC vaccine intradermally, or OC-L (2.5-5x106 oxidized tumor cells admixed with Montanide ISA 51 VG) 2-3 Days post T-cell infusion and on Day 16-18. Subjects will start receiving Bevacizumab at 15 mg/kg and vaccine (if available) starting Day 30 and every 3 weeks thereafter until end of study. (Funding Source - FDA OOPD)

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have received at least one vaccine under protocol UPCC-19809 or UPCC-29810.
* ECOG performance status 0 or 1.
* Subject has sufficient vaccine (2 vaccine doses are sufficient)
* Must be at least 4 weeks post-operative
* Blood coagulation parameters: PT such that international normalized ratio (INR) is less than1.5 (or an in-range INR, usually between 2 and 3, if a subject is on a stable dose of therapeutic warfarin for management of venous thrombosis including pulmonary thromboembolus) and a PTT less than1.2 times the upper limit of normal.
* Subject must be 18 years of age or older.
* Life expectancy of greater than 4 months.
* Normal organ and bone marrow function as defined by: Absolute neutrophil count greater than 1,000/microliter, Platelets greater than 100,000/microliter, Hematocrit greater than 30%, AST (SGOT)/ALT(SGPT) less than 2.5 X institutional upper limit of normal, Bilirubin less than 2.0 mg/dL unless secondary to bile duct blockage by tumor, and Creatinine less than 1.8 mg/dL

Exclusion Criteria:

* Subjects who require or are likely to require more than a two-week course of corticosteroids for intercurrent illness. Subjects must complete therapy prior to enrollment. Topical corticosteroids should be stopped at least 2 weeks prior to enrollment and systemic corticosteroids should be stopped at least 4 weeks prior to enrollment.
* Subjects with any acute infection that requires specific therapy. Acute therapy must have been completed at least seven days prior to study enrollment
* Subjects with any underlying conditions, which would contraindicate therapy with, study treatment (or allergies to reagents used in this study).
* Subjects with prior history or symptoms suggestive of partial or complete bowel obstruction.
* Subjects receiving class III antiarrythmic medications.
* Subjects receiving medications that might affect immune function. Additionally, H2 blockers are excluded, as are all antihistamines five days before and five days after each injection of study drug. NOTE: The following are exceptions: Proton pump Inhibitors (PPIs), NSAIDS including COX-2 inhibitors, acetaminophen.
* Subjects who are allergic to Aspirin are excluded
* Development of clinically significant co morbid disease that would contraindicate study therapy or confuse interpretation of study results.
* Subjects with a History of bowel obstruction, including sub-occlusive disease, related to the underlying disease and history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess.
* Subjects with evidence of recto-sigmoid involvement by pelvic examination or bowel involvement on CT scan or clinical symptoms of bowel obstruction.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-03; Primary Completion 2015-10 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 5 Years
  Dose limiting toxicity is defined as the occurrence of treatment-related adverse events.

SECONDARY OUTCOMES:
Tumor response | 5 years
  Tumor response will be estimated by measures of tumor burden and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Janos Tanyi, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Bobisse S, Bianchi V, Tanyi JL, Sarivalasis A, Missiaglia E, Petremand R, Benedetti F, Torigian DA, Genolet R, Barras D, Michel A, Mastroyannis SA, Zsiros E, Dangaj Laniti D, Tsourti Z, Stevenson BJ, Iseli C, Levine BL, Speiser DE, Gfeller D, Bassani-Sternberg M, Powell DJ Jr, June CH, Dafni U, Kandalaft LE, Harari A, Coukos G. A phase 1 trial of adoptive transfer of vaccine-primed autologous circulating T cells in ovarian cancer. Nat Cancer. 2023 Oct;4(10):1410-1417. doi: 10.1038/s43018-023-00623-x. Epub 2023 Sep 21. PMID 37735588